CLINICAL TRIAL: NCT06751446
Title: Enhancing the Ability of Critical Thinking and Clinical Reasoning Among Nursing Students on Post-operative Management Through Scenario-Based Simulation
Brief Title: Improving Critical Thinking and Clinical Reasoning in Nursing Students Through Post-Operative Scenario-Based Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Sadia Sultana Tonny, Principal Investigator, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GCCN/IRB/2024-12
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Nursing Education; Teaching Method

STUDY DESIGN:
Intervention Model Description: Intervention Group Control Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scenario-Based Simulation Training (Experimental): Students allocated to the intervention group through block randomisation will participate in scenario-based simulation training. The Principal Investigator (PI) and GCCN faculty will guide the students using PI-developed videos and scenarios. The training will incorporate cases that depict abnormal signs and symptoms, fostering active learning and challenging students to apply practical skills. Later, students will engage in group-based skills training for repeated practice and reinforcement.
  Interventions: Other: Scenario-based Simulation Skill Training
- Traditional Skills Training (Experimental): Students allocated to the control group through block randomisation will undergo traditional skills training. The Principal Investigator (PI) and GCCN faculty will demonstrate and train them in postoperative nursing management techniques. Later, students will practice independently in a skills lab under the guidance of the PI and GCCN faculty. Finally, all students will participate in a skills evaluation and knowledge post-test and provide free comments. To address potential ethical concerns, after the study's completion, the PI and GCCN faculty will provide the control group with training in scenario-based simulation and show them the developed videos on post-operative nursing management.
  Interventions: Other: Traditional Skill Training

INTERVENTIONS:
Other: Scenario-based Simulation Skill Training — Scenario-based simulation is an educational approach that immerses students in realistic clinical scenarios, allowing them to practice decision-making and problem-solving in a safe, controlled environment. It challenges students to assess patient data, identify priorities, and implement interventions. Through guided debriefing sessions, students reflect on their actions, justify their decisions, and explore alternative strategies.
  Arms: Scenario-Based Simulation Training
Other: Traditional Skill Training — Traditional skill training in nursing education focuses on developing core technical skills through direct instruction, demonstrations, and hands-on practice. It emphasises mastery of essential tasks and conducting patient assessments. Students follow standardized protocols and procedures to ensure patient safety and accuracy in their practice
  Arms: Traditional Skills Training

SUMMARY:
The goal of this clinical trial is to determine whether scenario-based simulation training can effectively enhance critical thinking and clinical reasoning skills in nursing students in Bangladesh, focusing on postoperative nursing management.

The main questions it aims to answer are:

1. Does scenario-based simulation training improve critical thinking and clinical reasoning skills in postoperative nursing management?
2. Is scenario-based simulation training more effective than traditional skills training in enhancing these skills?

Researchers will compare an intervention group (receiving scenario-based simulation training) to a control group (receiving traditional skills training) to see if the intervention leads to greater improvements in critical thinking and clinical reasoning abilities.

Participants will:

* Attend lectures on postoperative nursing care, take a pre-test, and be randomly assigned to either the intervention or control group.
* The intervention group will undergo scenario-based simulation training, while the control group will receive traditional skills training.
* Both groups will engage in individual practice and complete post-training evaluations to assess critical thinking, clinical reasoning, and overall competency

This study aims to identify an effective teaching strategy for nursing students, enhancing their ability to handle complex clinical situations and improving patient care quality.

DETAILED DESCRIPTION:
This study, titled "Enhancing the Ability of Critical Thinking and Clinical Reasoning among Nursing Students on Post-operative Management through Scenario-Based Simulation," evaluates the impact of scenario-based simulation training on developing critical thinking and clinical reasoning skills in 2nd-year Bachelor of Science in Nursing (BSN) students at the Grameen Caledonian College of Nursing (GCCN), Bangladesh.

Design and Methodology:

The research employs a prospective, open-label, randomised controlled trial (RCT) with a 1:1 parallel design and block randomization. The study consists of 57 participants, split into an intervention group (scenario-based simulation training) and a control group (traditional skills training).

* Study Duration: 11 months from November 2024 to September 2025, including preparation, intervention (3 months), and analysis.
* Educational Context: Participants will have no prior exposure to postoperative nursing theory or practice before this intervention.

Intervention Protocol

1. One week ( Both for intervention group and control group)

   * Two lectures on postoperative nursing management, critical thinking, and clinical reasoning.
   * Pre-test to assess baseline knowledge and randomise participants.
2. One to two weeks ( Based on the school schedule)

Training:

* Intervention Group: scenario-based simulation, including group activities with realistic clinical cases, guided debriefing, and individual practice.
* Control Group: Traditional skills training with standard demonstrations and hands-on practice.

Independent Practice:

• Individual practice in skill labs to reinforce learning.

Evaluation:

* Skills and knowledge assessments using a standardised checklist and post-tests.
* Participant reflections were collected for qualitative insights.

Evaluation Metrics

Primary Outcome:

Development of critical thinking and clinical reasoning, assessed using a customised checklist that evaluates domains such as analysis, inference, and evaluation.

Secondary Outcomes:

* Knowledge improvement through pre- and post-tests.
* Practical skills in postoperative management.
* Qualitative insights from participant reflections.

Technical Aspects

Randomisation:

Block randomisation is based on pre-test scores, ensuring balanced baseline knowledge across groups.

Assessment Tools:

* Knowledge Test: A 25-item multiple-choice questionnaire assessing theoretical understanding.
* Critical Thinking and Clinical Reasoning Checklist: Developed based on a theoretical framework by Facione and validated by Hiroshima University nursing faculty.
* Skills Evaluation: Measures ability in critical and practical components of postoperative nursing care.

Ethical and Data Management

* Ethical approval is secured from GCCN's Institutional Review Board (IRB).
* Participants' data are anonymised, securely stored on a cloud system, and will be deleted after five years.
* Participation is voluntary, with informed consent required, and withdrawal allowed without penalties.

Significance This study addresses skill gaps in critical thinking and clinical reasoning among Bangladeshi nursing students. Findings will inform curriculum improvements and promote innovative teaching strategies, with broader implications for global nursing education.

ELIGIBILITY:
Inclusion Criteria:

* 2nd-year BSN students at GCCN who take "Adult medical & surgical nursing."
* Students who provide informed consent to participate in the study.

Exclusion Criteria:

•Students who have completed theory class and clinical practice in the postoperative ward in any hospital.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Ability of critical thinking and clinical reasoning with skill | 6-7 weeks after baseline data collection
  The primary outcome, critical thinking and clinical reasoning skills, will be assessed using a validated checklist covering five domains: analysis, inference, evaluation, inductive reasoning, and deductive reasoning. Students' performance in simulations or traditional skill demonstrations will be scored based on practical skills, critical thinking, and clinical reasoning. Trained evaluators will observe and score students' ability to identify patient problems, make evidence-based decisions, and explain their reasoning during debriefing sessions, ensuring a comprehensive assessment of these skills.The postoperative skill evaluation checklist includes practical skills, critical thinking, and clinical reasoning. The overall total score is 100: 48 for postoperative skill, 32 for critical thinking ability, and 20 for clinical reasoning ability. This ranges from 0 - 100. Higher scores show higher skill & ability, and lower score indicates less skill and ability.

SECONDARY OUTCOMES:
Critical Thinking Ability | 6-7 weeks after baseline data collection
  PI and the supervisor developed a questionnaire based on the theoretical model. Total score ranges from 0-32. A higher score shows higher ability, and a lower score indicates less ability.
Clinical Reasoning Ability | 6-7 weeks after baseline data collection
  PI and the supervisor developed a questionnaire based on the theoretical model.Total score ranges from 0-20. A higher score shows higher ability, and a lower score indicates less ability.
Post Operative Management Skill | 6-7 weeks after baseline data collection
  It was adapted from a questionnaire from the adult medical and surgical nursing department of Hiroshima University. The postoperative skill score ranges from 0 to 48. Higher scores show higher skill, and a lower score indicates less skill.
Knowledge Test Score | 1 week after lecture session and 6-7 week after baseline data collection
  PI and the supervisor developed a questionnaire based on the medical & surgical nursing textbooks.The test will have a total score range of 0-25. A higher score indicates a higher level of knowledge, whereas a lower score indicates a lesser level of knowledge.
Free Commnents | 6-7 weeks after baseline data collection
  The researcher developed a questionnaire. It has five comments.Free comments will undergo thematic analysis to identify key themes and patterns, with results presented as a narrative summary using illustrative quotes or making categories to describe their responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Grameen Caledonian College of Nursing, Dhaka, Turag, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Share according to request to the PI and Supervisor
Time Frame: 2025 - 2026
Access Criteria: sadiasultana43329@gmail.com